CLINICAL TRIAL: NCT05062902
Title: An Novel Medical System for Quantitative Diagnosis and Personalized Precision Botulinum Neurotoxin Injection in Chronic Pelvic Pain Management
Brief Title: A Novel Medical System for Quantitative Diagnosis and Personalized Precision Botulinum Neurotoxin Injection in Chronic Pelvic Pain Management
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: HillMed Inc. (Industry)
Collaborators: Baylor College of Medicine (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Nicholas Dias, Principal Research Scientist, HillMed Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R44HD107822 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-09-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Cystitis; Chronic Pain; Pelvic Floor; Relaxation; Pelvic Floor Disorders
Keywords: hypertonicity; chronic pelvic pain; electromyography
MeSH Terms: conditions — Cystitis, Interstitial; Chronic Pain; Pelvic Floor Disorders; Muscle Hypertonia | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Template Injection (Active Comparator): For the standard template injection, 200 units of BoNT diluted in 6mL of preservative saline will be prepared. 1/4 of the prepared BoNT solution will be administered to each of the pubococcygeus and puborectalis muscle at 5 and 7 o'clock position, respectively. The index finger will be used for palpation as the 20-gauge spinal needle with a trumpet guide (i.e. paracervical block kit) piercing through the vaginal mucosa to the intended muscle groups. The syringe will be withdrawn before each injection to avoid intravascular injection.
  Interventions: Drug: Botulinum Neurotoxin
- Guided Injection (Experimental): For the guided injection, pelvic floor injections (total of 4) will be made to the pubococcygeus and puborectalis muscles each, at NMJ locations (1.5 ml per site), at patient-specific locations and depths identified from vaginal HD-sEMG recordings. NMJ mappings will be generated for each participant. The channel locations will provide angle measurements for each NMJ. The device will calculate these parameters based on acquired HD-sEMG. The index finger will be used for palpation and guidance of injection needle through the vaginal mucosa to the defined injection sites. The BoNT dosage with respect to the total 200 units administered to each site will be patient specific, determined as the ratio of the resting average resting root-mean square (RMS) value of a specific region divided by the total average resting RMS.
  Interventions: Device: High Density Surface Electromyographic, precision botulinum neurotoxin injection guidance medical device; Drug: Botulinum Neurotoxin

INTERVENTIONS:
Device: High Density Surface Electromyographic, precision botulinum neurotoxin injection guidance medical device — A personalized, precision botulinum neurotoxin injection guidance medical device, utilizing an intra-vaginal high-density surface EMG system to optimize the treatment outcomes in chronic pelvic pain (CPP) management.
  Arms: Guided Injection
Drug: Botulinum Neurotoxin — Botulinum neurotoxin will be injected into the pelvic floor muscles following either a standard template (standard injection arm), or guided using high-density surface EMG (guided arm).

SUMMARY:
The purpose of this study is to evaluate if it is possible to use intravaginal high-density surface electromyography to guide Botulinum neurotoxin (BoNT) injection to treat pelvic floor muscle overactivity that complicates Chronic Pelvic Pain (CPP).

DETAILED DESCRIPTION:
The management of pelvic floor overactivity (PFOA) using focal BoNT injection has been gaining clinical interest. Evidence has shown that BoNT injections to the levator ani in patients with CPP generated a greater than 50% improvement in symptoms at least 72% of the time, suggesting a promising efficacy of BoNT therapy. The current clinical standard for BoNT injection employs a fixed injection template or the manual palpation of a contracted muscle, followed by an injection towards the palpating finger. As such, the injection is highly subjective, operator-dependent, variable, and not tailored to individual patients, which may lead to inconsistent outcomes. Trigger point targeted injections have been practiced for many years worldwide, yet a recent randomized controlled trial reported no significant difference in outcome between trigger point targeted BoNT injections versus a saline placebo. Furthermore, it has also been reported that neuromuscular junction (NMJ) and trigger points are distributed in well-defined separate areas with a distance of approximately 10 mm apart. It has also been shown that BoNT injections made 10 mm away from the NMJ can reduce the efficacy of BoNT by 46%. Therefore, injections targeted at the trigger point may, in turn, compromise therapeutic efficacy.

The rationale of this study is that BoNT acts at the NMJ, where the neuromuscular junctions are densely located. By specifying the muscle(s) responsible for the pelvic floor overactivity, and the offending NMJ using high density surface electromyography (HD-sEMG), BoNT can be injected with greater accuracy and objectivity to optimize treatment efficacy. The investigators aim to test the hypothesis that interstitial cystitis patients in the guided injection arm will demonstrate lower hypertonic metrics and improved quality of life. The purpose of this study is to provide preliminary evidence supporting the use of HD-sEMG and NMJ mapping to guide BoNT efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for interstitial cystitis/bladder pain syndrome (IC/BPS) patients will be:

  1. Woman aged 18 to 60.
  2. Have a clinical diagnosis of IC/BPS.
  3. Pain, pressure, or discomfort in the bladder and/or pelvic area for the past 6 months or more, associated with lower urinary tract symptoms (such as frequency of urination), in the absence of other explanation of the symptoms (e.g., urinary tract infection).
  4. Myofascial pain diagnosed with palpable contracted muscle fibers.
  5. Pelvic muscle tenderness by assessment of pelvic floor muscles on digital pelvic examination.
  6. Pelvic floor hypertonicity (PFH), measured using vaginal manometry (pressure > 35 cm∙H2O).
  7. Ability to provide informed consent.

Exclusion Criteria:

* Exclusion criteria consist of the following:

  1. History of pelvic malignancy and sexually transmitted diseases.
  2. Bleeding disorder such as coagulopathy
  3. History of neurological disorders, such as spinal cord injury, multiple sclerosis, amyotrophic lateral sclerosis or myasthenia gravis.
  4. Pregnancy, breast feeding or desiring for pregnancy in the coming year.
  5. Subjects with history of pelvic surgery (e.g., pain from mid-urethral sling or pelvic mesh),
  6. Pelvic malignancy (urinary tract, gynecologic, gastrointestinal)
  7. Active fistula
  8. Radiation cystitis
  9. Cyclophosphamide cystitis
  10. Pre-existing anorectal disorders
  11. Infections near the injection sites
  12. History of drug or alcohol abuse
  13. Hypersensitivity to BoNT
  14. Steroids or hormone usage will be carefully considered by the research team for inclusion.

Participants with on-going BoNT therapies will not be screened until the complete drug washout is confirmed.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hypertonic metrics of the pelvic muscles defined by intra-vaginal surface EMG | Baseline
  The pelvic floor hypertonicity will be assessed by evaluating the amplitudes of intra-vaginal high-density surface electromyography recordings.
Hypertonic metrics of the pelvic muscles defined by intra-vaginal surface EMG | 1-Month Post Injection
  The pelvic floor hypertonicity will be assessed by evaluating the amplitudes of intra-vaginal high-density surface electromyography recordings.
Hypertonic metrics of the pelvic muscles defined by intra-vaginal surface EMG | 3-Months Post Injection
  The pelvic floor hypertonicity will be assessed by evaluating the amplitudes of intra-vaginal high-density surface electromyography recordings.

SECONDARY OUTCOMES:
Global response assessment | 1-Month Post Injection
  Compared to prior to the treatment, is the patient very much better, much better, a little better, no change, a little worse, much worse, or very much worse.
Global response assessment | 3-Months Post Injection
  Compared to prior to the treatment, is the patient very much better, much better, a little better, no change, a little worse, much worse, or very much worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided